CLINICAL TRIAL: NCT02859415
Title: Phase I/II Evaluation of Continuous 24h Intravenous Infusion of Mithramycin, an Inhibitor of Cancer Stem Cell Signaling, in Patients With Primary Thoracic Malignancies or Carcinomas, Sarcomas or Germ Cell Neoplasms With Pleuropulmonary Metastases
Brief Title: Continuous 24h Intravenous Infusion of Mithramycin, an Inhibitor of Cancer Stem Cell Signaling, in People With Primary Thoracic Malignancies or Carcinomas, Sarcomas or Germ Cell Neoplasms With Pleuropulmonary Metastases
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow/Insufficient accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Schrump, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160152; 16-C-0152
Record Dates: First submitted 2016-08-06; First posted 2016-08-09 (Estimated); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Esophageal Neoplasms; Lung Neoplasms; Mesothelioma; Thymus Neoplasms; Neoplasms, Germ Cell and Embryonal
Keywords: Metastatic Colorectal Cancer; Sarcoma; ABCB4 Liver Toxicity; ABCB11 Hepatotoxicity; Metastatic Renal Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms; Mesothelioma; Thymus Neoplasms; Neoplasms, Germ Cell and Embryonal; Colorectal Neoplasms; Sarcoma; Kidney Neoplasms | interventions — Plicamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I/Escalating doses of Mithramycin (Experimental): Escalating doses of Mithramycin
  Interventions: Drug: Mithramycin
- Phase II/Mithramycin administered at Maximum Tolerated Dose (MTD) (Experimental): Mithramycin administered at MTD
  Interventions: Drug: Mithramycin

INTERVENTIONS:
Drug: Mithramycin — Phase 1: 24 hour intravenous infusion of mithramycin given once every 14 days at escalating doses; Phase 2: 24 hour intravenous infusion of mithramycin given once every 14 days at MTD established in phase 1
  Other Names: Plicamycin

SUMMARY:
Background:

Mithramycin is a new cancer drug. In another study, people with chest cancer took the drug 6 hours a day for 7 straight days. Many of them had liver damage as a side effect. It was discovered that only people with certain genes got this side effect. Researchers want to test mithramycin in people who do not have those certain genes.

Objectives:

To find the highest safe dose of mithramycin that can be given to people with chest cancer who have certain genes over 24 hours instead of spread out over a longer period of time. To see if mithramycin given as a 24-hour infusion shrinks tumors.

Eligibility:

People ages 18 and older who have chest cancer that is not shrinking with known therapies, and whose genes will limit the chance of liver damage from mithramycin

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood and urine tests
* Lung and heart function tests
* X-rays or scans of their tumor
* Liver ultrasound
* Tumor biopsy
* Participants will be admitted to the hospital overnight. A small plastic tube (catheter) will be inserted in the arm or chest. They will get mithramycin through the catheter over about 24 hours.
* If they do not have bad side effects or their cancer does not worsen, they can repeat the treatment every 14 days.
* Participants will have multiple visits for each treatment cycle. These include repeats of certain screening tests.
* After stopping treatment, participants will have weekly visits until they recover from any side effects.

DETAILED DESCRIPTION:
Background:

Increasing evidence indicates that activation of stem cell gene expression is a common mechanism by which environmental carcinogens mediate initiation and progression of thoracic malignancies. Similar mechanisms appear to contribute to extra-thoracic malignancies that metastasize to the chest. Utilization of pharmacologic agents, which target gene regulatory networks mediating "stemness" may be novel strategies for treatment of these neoplasms. Recent studies performed in the Thoracic Epigenetics

Laboratory, National Cancer Institute (NCI), demonstrate that under exposure conditions potentially achievable in clinical settings, mithramycin diminishes stem cell gene expression and markedly inhibits growth of lung and esophageal cancer and malignant pleural mesothelioma (MPM) cells in vitro and in vivo. These findings add to other recent preclinical studies demonstrating impressive anti-tumor activity of mithramycin in epithelial malignancies and sarcomas that frequently metastasize to the thorax.

Primary Objectives:

* Phase I component: To determine pharmacokinetics, toxicities, and maximum tolerated dose (MTD) of mithramycin administered as a continuous 24h infusion in patients with primary thoracic malignancies or carcinomas, sarcomas or germ cell tumors metastatic to the chest.
* Phase II component: To determine objective response rates (Complete Response (CR) + Partial Response (PR) of mithramycin administered as 24h intravenous infusions in patients with primary thoracic malignancies or carcinomas, sarcomas or germ cell tumors metastatic to the chest.

Eligibility:

* Patients with measurable inoperable, histologically confirmed lung and esophageal carcinomas, thymic neoplasms, germ cell tumors, malignant pleural mesotheliomas or chest wall sarcomas, as well as patients with gastric, colorectal or renal cancers and sarcomas metastatic to the thorax are eligible.
* Patients with favorable germline single nucleotide polymorphisms (SNPs) in ATP Binding Cassette Subfamily B Member 4 (ABCB4), ATP Binding Cassette Subfamily B Member 11 (ABCB11), Ral binding protein (RALBP) or Cytochrome P450 Family 8 Subfamily B Member 1 (CYP8B1) that are associated with resistance to mithramycin-induced hepatotoxicity.
* Patients must have had or refused first-line standard therapy for their malignancies.
* Patients must be 18 years or older with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2, without evidence of unstable or decompensated myocardial disease. Patients must have adequate pulmonary reserve evidenced by forced expiratory volume (FEV1) and diffusing capacity for carbon monoxide (DLCO) equal to or greater than 30% predicted; Oxygen saturation >= 92% on room air. ABG will be drawn if clinically indicated.
* Patients must have a platelet count greater than or equal to 100,000, an absolute neutrophil count (ANC) equal to or greater than 1500 without transfusion or cytokine support, a normal prothrombin time (PT)/partial thromboplastin time (PTT), and adequate hepatic function as evidenced by a total bilirubin of < 1.5 x upper limits of normal (ULN) and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) <= 3 X ULN.
* Serum creatinine within normal institutional limits or creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.

Design:

* Single arm Phase I dose escalation to define pharmacokinetics, toxicities and maximum tolerated dose (MTD).
* Patient cohorts will receive 24hour(h) infusions of mithramycin targeting total doses previously administered during 7 daily six hour infusions at 30-50 mcg/kg.
* The 24h infusions will be administered every 14 days (1 cycle). Four cycles will constitute one course of therapy.
* Pharmacokinetics and toxicity assessment to define MTD will be assessed during Cycle 1 of the first course of therapy.
* Due to uncertainties regarding potential cumulative toxicities, no intra-patient dose escalation will be allowed.
* Once MTD has been defined, patients will be enrolled into two cohorts (primary thoracic malignancy vs neoplasm of non-thoracic origin metastatic to the chest) to determine clinical response rates at the MTD, using a Simon Optimal Two Stage Design for Phase II Clinical Trials targeting an objective response rate (Response Evaluation Criteria in Solid Tumors (RECIST) of 30%.
* Following each course of therapy, patients will undergo restaging studies. Patients exhibiting objective response to therapy or stable disease by RECIST criteria will be offered an additional course of therapy.
* Patients exhibiting disease progression will be removed from study.
* Biopsies of index lesions will be obtained at baseline and on Day 4 of the first cycle of therapy for analysis of pharmacodynamic endpoints. Optional tumor biopsies may be requested at the completion of Course 1 (4 cycles) and in patients exhibiting objective responses.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with measurable inoperable, histologically confirmed non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), esophageal carcinomas, thymic neoplasms, germ cell tumors, malignant pleural mesotheliomas or chest wall sarcomas, as well as patients with gastric, colorectal, pancreas or renal cancers, and sarcomas metastatic to thorax.
* Histologic confirmation of disease in the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI), National Institutes of Health (NIH).
* Disease amenable to biopsy via percutaneous approach or other minimally invasive procedures such as thoracoscopy, bronchoscopy, laparoscopy, or gastrointestinal (GI) endoscopy.
* Age >= 18.
* Eastern Cooperative Oncology Group (ECOG) status 0-2.
* Patients must have had, or refused first-line standard chemotherapy for their inoperable malignancies.
* Patients must have had no chemotherapy, biologic therapy, or radiation therapy for their malignancy for at least 30 days prior to treatment. Patients may have received localized radiation therapy to non-target lesions provided that the radiotherapy is completed 14 days prior to commencing therapy, and the patient has recovered from any toxicity. At least 3 half-lives must have elapsed since monoclonal antibody treatment. At least 6 weeks must have elapsed between mitomycin C or nitrosourea treatment.
* Patients must have adequate organ and marrow function as defined below:

  1. Hematologic and Coagulation Parameters

     * Peripheral absolute neutrophil count (ANC) greater than or equal to 1500/mm(3)
     * Platelets greater than or equal to 100,000/ mm(3) (transfusion independent)
     * Hemoglobin greater than or equal to 8 g/dL (PRBC transfusions permitted)
     * Prothrombin Time (PT)/partial thromboplastin time (PTT) within normal limits (patient may be eligible for trial if abnormality is deemed clinically insignificant and cleared for protocol therapy by Hematology Consult service)
  2. Hepatic Function

     * Bilirubin (total) < 1.5 times upper limit of normal (ULN)
     * Alanine aminotransferase (ALT) Serum glutamic pyruvic transaminase(SGPT) less than or equal to 3.0 times ULN
     * Albumin > 2 g/dL
  3. Renal Function

     * Creatinine within normal institutional limits or creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
     * Normal ionized calcium, magnesium and phosphorus (can be on oral supplementation)
* Cardiac Function: Left ventricular ejection fraction (EF) >40% by echocardiogram, multigated acquisition scan (MUGA), or cardiac magnetic resonance (MR).
* Ability of subject to understand, and be willing to sign informed consent.
* Female and male patients (and when relevant their partners) must be willing to practice birth control (including abstinence) during and for 2 months after treatment if female of childbearing potential or male having sexual contact with a female of childbearing potential.
* Patients must be willing to undergo 2 tumor biopsies.

EXCLUSION CRITERIA:

* Patients with unfavorable ATP Binding Cassette Subfamily B Member 4 (ABCB11), Ral binding protein (RALBP) or Cytochrome P450 Family 8 Subfamily B Member 1 (CYP8B1) genotypes associated with mithramycin-mediated hepatotoxicity
* Clinically significant systemic illness (e.g. serious active infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the judgment of the PI would compromise the patient's ability to tolerate protocol therapy or significantly increase the risk of complications.
* Patients with cerebral metastases.
* Patients with any of the following pulmonary function abnormalities will be excluded: forced expiratory volume (FEV), < 30% predicted; diffusing capacity for carbon monoxide (DLCO), < 30% predicted (post-bronchodilator); Oxygen saturation less than or equal to 92% on room air (per vital sign measurement). Arterial blood gas will be drawn if clinically indicated.
* Patients with evidence of active bleeding, intratumoral hemorrhage or history of bleeding diatheses, unless specifically occurring as an isolated incident during reversible chemotherapy-induced thrombocytopenia.
* Patients on therapeutic anticoagulation. Note: Prophylactic anticoagulation (i.e. intraluminal heparin) for venous or arterial access devices is allowed.
* Patients who are concurrently receiving or requiring any of the following agents, which may increase the risk for mithramycin related toxicities, such as hemorrhage:

  * Thrombolytic agents
  * Aspirin or salicylate-containing products, which may increase risk of hemorrhage
  * Dextran
  * Dipyridamole
  * Sulfinpyrazone
  * Valproic acid
  * Clopidogrel
* Lactating or pregnant females (due to risk to fetus or newborn, and lack of testing for excretion in breast milk).
* Patients with history of human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) due to potentially increased risk of mithramycin toxicity in this population.
* Hypersensitivity to mithramycin.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-C-0152.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated for slow/insufficient accrual before reaching phase II.
Groups:
- Phase I Dose Level 1 Mithramycin 60 mcg/kg: Phase I Dose Level 1 Mithramycin 60 mcg/kg
  Mithramycin: Phase 1: 24 hour intravenous infusion of mithramycin given once every 14 days at escalating doses..
- Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg: Phase I Dose Level -1 Mithramycin 60 mcg/kg followed by Mithramycin 30 mcg/kg
  Mithramycin: Phase 1: 24 hour intravenous infusion of mithramycin given once every 14 days at escalating doses.
Period: Overall Study
Arm/Group | Phase I Dose Level 1 Mithramycin 60 mcg/kg | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg
Started | 1 | 2
Completed | 0 | 1
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Off treatment due to cardiac event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 1 Mithramycin 60 mcg/kg | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (0) | 49.35 (18.88) | 52.33 (14.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD is defined as the number of participants experiencing a dose-limiting toxicity (DLT). A DLT is defined as Grade 4 or greater anemia or neutropenia exceeding 5 days duration, thrombocytopenia requiring transfusion, or Grade 3 or greater nonhematologic toxicity possibly, probably, or definitely related to the investigational therapy excluding alopecia during Cycle 1 of therapy.
Time Frame: At the end of first 14 day cycle at each dose level
Measure: Number; unit: mcg/kg
Groups:
- All Participants: All participants in phase I dose level 1 and dose level -1.
Arm/Group | All Participants
Number analyzed (Participants) | 3
mcg/kg | NA — The MTD was not found because we did not have enough participant participation.

2. Primary Outcome: Number of Participants Whose Best Response is a Complete Response (CR) or Partial Response (PR)
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: every 8 weeks until at disease progression, approximately 3.5 months
Population: One participant in the first group only received one dose, thus was not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 Mithramycin 60 mcg/kg | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg
Number analyzed (Participants) | 0 | 2
Participants
  Complete Response |  | 0
  Partial Response |  | 0

3. Secondary Outcome: To Ascertain if Mithramycin Inhibits Stem Cell Gene Expression in Participants With Thoracic Malignancies
Description: Studies on tumor tissue obtained during baseline /previous biopsy (if available), Cycle 1 Day 4(+/- 3 days), and possible treatment evaluation following Course 1. Plasma and blood will also be collected.
Time Frame: baseline, Cycle 1 Day 4 (+/- 3 days), and possible treatment evaluation following Course 1
Population: No data was collected thus this outcome measure was not done.
Arm/Group | Phase I Dose Level 1 Mithramycin 60 mcg/kg | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Evaluate Gene Expression, Deoxyribonucleic Acid (DNA) Methylation and Micro-ribonucleic Acid (RNA) Profiles in Pre- and Post-treatment Tumor Biopsies
Description: Studies on tumor tissue obtained during baseline /previous biopsy (if available), Cycle 1 Day 4(+/- 3 days), and possible treatment evaluation following Course 1.
Time Frame: baseline, Cycle 1 Day 4 (+/- 3 days), and possible treatment evaluation following Course 1
Population: No data was collected thus this outcome measure was not done.
Arm/Group | Phase I Dose Level 1 Mithramycin 60 mcg/kg | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: To Compare Gene Expression, Deoxyribonucleic Acid (DNA) Methylation and Micro-ribonucleic Acid (RNA) Profiles in Participant Tumor Biopsies With Treatment Response Profiles in Pre-clinical Studies
Description: as for outcome 4
Time Frame: baseline, Cycle 1 Day 4 (+/- 3 days), and possible treatment evaluation following Course 1
Population: No data was collected thus this outcome measure was not done.
Arm/Group | Phase I Dose Level 1 Mithramycin 60 mcg/kg | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: To Examine if Mithramycin Decreases Pluripotent Cancer Stem Cells (Side Population)
Description: as for outcome 4
Time Frame: baseline, Cycle 1 Day 4 (+/- 3 days), and possible treatment evaluation following Course 1
Population: No data was collected thus this outcome measure was not done.
Arm/Group | Phase I Dose Level 1 Mithramycin 60 mcg/kg | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: To Develop Methodologies for Assessing Effects of Mithramycin on Cancer Stem Cells, Hematopoietic Stem Cells, Mesenchymal Stem Cells, and Circulating Tumor Cells (CTC)
Description: as for outcome 3
Time Frame: baseline, Cycle 1 Day 4 (+/- 3 days), and possible treatment evaluation following Course 1
Population: No data was collected thus this outcome measure was not done.
Arm/Group | Phase I Dose Level 1 Mithramycin 60 mcg/kg | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 1 month and 4 days, and 3 months and 17 days for the first and second group respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 Mithramycin 60 mcg/kg | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

9. Other Pre Specified Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: A DLT is defined as Grade 4 or greater anemia or neutropenia exceeding 5 days duration, thrombocytopenia requiring transfusion, or Grade 3 or greater nonhematologic toxicity possibly, probably, or definitely related to the investigational therapy excluding alopecia during Cycle 1 of therapy.
Time Frame: Cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 Mithramycin 60 mcg/kg | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 1 month and 4 days, and 3 months and 17 days for the first and second group respectively.
Arm/Group | Phase I Dose Level 1 Mithramycin 60 mcg/kg | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 1 Mithramycin 60 mcg/kg (N=1) | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg (N=2)
Alanine aminotransferase (Investigations) | 0 (0) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 1 Mithramycin 60 mcg/kg (N=1) | Phase I Dose Level -1 Mithramycin 60 mcg/kg Followed by Mithramycin 30 mcg/kg (N=2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (4)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (19)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (3)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (8)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT02859415/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT02859415/ICF_001.pdf